CLINICAL TRIAL: NCT01318876
Title: Active Surveillance of Adverse Events Following Immunization Among Healthcare Workers Immunized With the Influenza Vaccine
Brief Title: Surveillance for Adverse Events Following Influenza Immunization
Status: Completed | Type: Observational
Sponsor: PHAC/CIHR Influenza Research Network (Other Government)
Collaborators: GlaxoSmithKline (Industry); Institut National en Santé Publique du Québec (Other); Laval University (Other); CHU de Quebec-Universite Laval (Other); Mount Sinai Hospital, Canada (Other); IWK Health Centre (Other); Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other); The Ottawa Hospital (Other); University of British Columbia (Other)
Responsible Party: Principal Investigator, Gaston De Serres, Epidemiologist at the National Institute of Public Health of Quebec and professor of epidemiology at the University Laval, PHAC/CIHR Influenza Research Network
Other Study IDs: pcirn-surveillancehcw-1011
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Results first posted 2012-08-14 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Influenza; Vaccines Adverse Reaction
Keywords: influenza; vaccine safety; adverse events; health care workers
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- BC Children's and Women's Hospital, Vancouver.
- University of British Columbia, Vancouver.
- Health care workers in Halifax
- Health care workers from CHUQ hospitals
- Health care workers from Toronto
- Centre hospitalier et universitaire de Sherbrooke
- The Ottawa General Hospital, Ottawa

SUMMARY:
Influenza vaccines are continuously modified to adjust to the virus antigenic shifts or drifts, and its safety profile may vary. While generally considered safe, influenza vaccines have been associated in the past with increases in cases of Guillain-Barré syndrome (1976) and with oculorespiratory syndrome in 2001. Last year, with the vaccination against the pH1N1, an increase of allergic-like reactions was observed.

Passive surveillance is collecting notifications of adverse events (AE) on the whole population but the sensitivity of this system is not high and its timeliness is not necessarily optimal. Last year, with the new pandemic Influenza vaccine the investigators piloted a web-based active surveillance of a large number of health care workers (HCW) vaccinated with the new adjuvanted monovalent pH1N1 influenza vaccine (Arepanrix® GSK, Canada). Because healthcare workers (HCW) constituted a well-defined group with general good health and received the Influenza vaccine in priority, this group of people was well suited for monitoring the safety of the influenza vaccine. For this study, 6242 HCW were recruited in three different sites (5183 were from Quebec). A total of 468 events (local reactions, fever, systemic reactions, gastrointestinal and respiratory problems) were reported by 430 HCW. 80% of the HCW recruited completed at least one of the three surveys and 52% responded to all questionnaires. During this surveillance, the investigators didn't have unexpected findings but this active surveillance of adverse events among healthcare workers would have been effective enough to rapidly detect adverse events occurring at a rate ≥ 1 per 200 vaccinees. For this year the investigators want to expand the surveillance to more sites and more participants to be able to detect AE occurring at rates ≥ 1 per 500 vaccinees, and to increase the response rate to all three surveys in participants.

The main objective of this project is to estimate in HCW vaccinated against influenza the frequency of adverse events of sufficient severity to cause work absenteeism or medical consultation.

This year the network will include 5 Canadian hospitals (Quebec City, Vancouver, Toronto, Halifax, + another one ) with a total enrollment of >10 000 HCW. This should allow us to detect AE occurring at a rate of ≥ 1 per 500 vaccinees.

ELIGIBILITY:
Inclusion Criteria:

* To be a healthcare worker from one of the seven Canadian Hospitals participating in the Public Health Agency of Canada/Canadian Institutes for Health Research-Influenza Research Network (PCIRN): Quebec City, Toronto, Halifax, Vancouver, Ottawa and Sherbrooke.
* To have been immunized with the influenza vaccine 2010
* To have an email address
* To be 18 years old and older
* To have sign the consent form

Exclusion Criteria:

* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The active surveillance was conducted in five Canadian hospitals participating in the Public Health Agency of Canada/Canadian Institutes for Health Research-Influenza Research Network (PCIRN): Quebec City, Toronto, Halifax, Vancouver (2 sites), Ottawa and Sherbrooke. Healthcare workers immunized in these institutions were offered to participate in a web-based active surveillance of vaccine safety.
Sampling Method: Probability Sample
Enrollment: 7645 (Actual)
Dates: Start 2010-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Canada (7):
  - BC Children's and Women's Hospital, Vancouver, Vancouver, British Columbia
  - University of British Columbia,, Vancouver, British Columbia
  - Canadian Center for Vaccinology, Halifax, Halifax, Nova Scotia
  - The Ottawa General Hospital,, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Toronto, Ontario
  - Centre Hospitalier Universitaire de Québec, Québec, Quebec
  - Centre Hospitalier et Universitaire de Sherbrooke, Sherbrooke, Quebec

REFERENCES:
- [Derived] De Serres G, Gariepy MC, Coleman B, Rouleau I, McNeil S, Benoit M, McGeer A, Ambrose A, Needham J, Bergeron C, Grenier C, Sleigh K, Kallos A, Ouakki M, Ouhoummane N, Stiver G, Valiquette L, McCarthy A, Bettinger J; PHAC-CIHR influenza Research Network (PCIRN). Short and long-term safety of the 2009 AS03-adjuvanted pandemic vaccine. PLoS One. 2012;7(7):e38563. doi: 10.1371/journal.pone.0038563. Epub 2012 Jul 3. PMID 22802929

RESULTS

PARTICIPANT FLOW:
Period: Day 8 Survey
Arm/Group | Health Care Workers
Started | 7645
Completed | 5825
Not Completed | 1820
Not completed — email address invalid | 96
Not completed — survey not completed-don't know why | 1724
Period: Day 29 Survey
Arm/Group | Health Care Workers
Started | 7549 (All participants with a valid e-mail, have received the second survey)
Completed | 5724
Not Completed | 1825
Not completed — survey not completed-don't know why | 1825

BASELINE CHARACTERISTICS:
Groups:
- Health Care Workers: HCW who had completed at least 1 survey (n=6269) and not the number of participants enrolled in the study.
Arm/Group | Health Care Workers
Number analyzed (Participants) | 6269
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | NA — participants under 18 years old were not recruted.
  Between 18 and 65 years | 6269
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41.77 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4639
  Male | 1630

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Experienced a New Health Problem or the Worsening of an Existing Health Condition That Resulted in a Medical Consultation
Time Frame: at day 8 and 29
Measure: Number; unit: participants
Arm/Group | HCW From All Sites
Number analyzed (Participants) | 6269
participants | 153

2. Primary Outcome: Number of Participants Who Had Experienced a New Health Problem or the Worsening of an Existing Health Condition That Resulted in Work Absenteeism.
Time Frame: day 8 and 29
Measure: Number; unit: participants
Arm/Group | HCW From All Sites
Number analyzed (Participants) | 6269
participants | 254

ADVERSE EVENTS:
Arm/Group | HCW From All Sites
Serious Adverse Events (participants affected / at risk) | 6/6269
Other Adverse Events (participants affected / at risk) | 0/6269
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HCW From All Sites (N=6269)
Spontaneous intracranial hypotension (Vascular disorders) | 1 (1)
kidney stone (Renal and urinary disorders) | 1 (1)
uterine fibroids (Reproductive system and breast disorders) | 1 (1)
anaphylactic shock to peanuts (Immune system disorders) | 1 (1)
allergic reaction (received epinephrine) (Immune system disorders) | 1 (1)
bilateral pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Only 70% answered the 2 surveys. We don't know why 30% didn't complete the 2 surveys (were they too sick or not motivated).We didn't have a group of comparable unvaccinated individuals (to estimate the risks attributable to the vaccine).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No